CLINICAL TRIAL: NCT06943443
Title: Evaluation of the Effects of Vitamin D Levels on Miniscrew-Assisted Rapid Palatal Expansion Treatment
Brief Title: Effect of Serum Vitamin D on MARPE Treatment Response
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, KAZIM KAAN YILDIZ, Principal Investigator/ Research Assistant, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025550
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Maxillary Transverse Deficiency Class I Malocclusion Vitamin D Deficiency Orthodontic Tooth Movement Adolescent Health
Keywords: Marpe
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group MARPE Treatment with Vitamin D Supplementation (Experimental): This group will receive Miniscrew-Assisted Rapid Palatal Expansion (MARPE) Treatment combined with Vitamin D supplementation. The patients in this group will undergo MARPE treatment for palatal expansion and receive Vitamin D supplementation according to the levels identified by their endocrinology evaluation at the beginning of the study. Vitamin D supplementation aims to optimize bone metabolism during the treatment process. Serum Vitamin D levels will be monitored before and after treatment to assess the effectiveness of supplementation in improving treatment outcomes.
  Interventions: Device: Miniscrew-Assisted Rapid Palatal Expansion (MARPE) Treatment
- Control Group MARPE Treatment without Vitamin D Supplementation (Active Comparator): Arm Description: This group will undergo Miniscrew-Assisted Rapid Palatal Expansion (MARPE) Treatment without any Vitamin D supplementation. The patients in this group will receive standard MARPE treatment for palatal expansion, and their serum Vitamin D levels will not be measured or supplemented during the study. The aim of this group is to serve as a comparison to evaluate the effects of Vitamin D supplementation in the experimental group.
  Interventions: Device: Miniscrew-Assisted Rapid Palatal Expansion (MARPE) Treatment

INTERVENTIONS:
Device: Miniscrew-Assisted Rapid Palatal Expansion (MARPE) Treatment — Vitamin D Supplementation: Vitamin D plays a crucial role in calcium absorption, bone health, immune system function, and cellular growth. It is primarily obtained through sunlight exposure, certain foods, and supplements. In the context of your study, Vitamin D supplementation will be used to improve the Vitamin D levels in patients undergoing Miniscrew-Assisted Rapid Palatal Expansion (MARPE) treatment.
  Key Points:
  Purpose: To correct Vitamin D deficiency, which may affect bone metabolism and orthodontic treatment outcomes.
  Administration: Vitamin D supplementation is typically provided in the form of oral tablets or soft gels, with a usual dosage of 800-2000 IU per day, depending on the individual's baseline levels.
  Measurement: Vitamin D levels will be measured at the beginning and end of treatment using 25-hydroxyvitamin D (25(OH)D tests to assess the effectiveness of supplementation.
  Effect on MARPE: Adequate Vitamin D levels may support better bone remodeling and healing, pote

SUMMARY:
A total of 30 patients are planned to be included in the study during the first half of 2025, who will apply to the clinic. In our clinical routine, approximately 30% of RME patients are treated using the MARPE method. The patients will be randomly assigned to two different groups. The first group will be referred to the Pediatric Endocrinology outpatient clinic at NEU Faculty of Medicine for vitamin D level measurements at the beginning of the treatment. The second group will proceed with treatment as usual, without vitamin D measurement. At the end of the treatment, vitamin D levels of all patients in both groups will be measured.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate the potential impact of serum vitamin D levels on the outcomes of Miniscrew-Assisted Rapid Palatal Expansion (MARPE) treatment in young adults aged 15-18 years. A total of 30 patients presenting with maxillary transverse deficiency will be recruited during the first half of 2025. Patients will be randomly allocated to two groups. The intervention group will undergo vitamin D level assessment at the beginning of treatment and receive supplementation if found deficient, while the control group will proceed without initial vitamin D evaluation.

Serum 25-hydroxyvitamin D [25(OH)D] levels will be measured at T1 and T2 timepoints. Intraoral scans will be performed using an Itero device to assess changes in intercanine and intermolar widths, and the data will be analyzed using the ORTHOCAD software. Pain levels will be recorded by the patients using a Visual Analog Scale (VAS) on specified days during the expansion phase. This study intends to determine whether baseline vitamin D status and subsequent supplementation can improve the biological response and clinical efficiency of MARPE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Class I malocclusion
* Presence of maxillary transverse deficiency
* Adolescents aged between 15 and 18 years
* No systemic diseases, cleft lip/palate, or speech disorders
* No history of prior orthodontic treatment
* Willingness to undergo serum vitamin D testing
* Voluntary participation in the study with signed informed consent
* Good oral hygiene status

Exclusion Criteria:

* Patients with systemic diseases
* Patients who smoke
* Patients with poor oral hygiene
* Patients with cooperation or compliance issues
* Patients with intellectual disabilities
* Patients with unmonitored or insufficient pre-treatment vitamin D levels, including:
* Those who had insufficient vitamin D levels before treatment, were started on supplementation by the endocrinology department, but still had insufficient levels at the T2 measurement
* Those who were not tested before treatment but were found to have sufficient vitamin D levels only at T2

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in Intermolar and Intercanine Widths After MARPE Treatment | At baseline (T1) and after expansion phase (T2), approximately 6 weeks apart
  Intermolar and intercanine width changes will be assessed using intraoral digital scans obtained with an iTero scanner. The width measurements will be made using ORTHOCAD software to determine the amount of skeletal expansion achieved with MARPE treatment.

SECONDARY OUTCOMES:
Change in Serum Vitamin D Levels | Baseline (T1) and Post-treatment at Week 8 (T2)
  Serum 25-hydroxyvitamin D [25(OH)D] levels will be measured in both groups. The intervention group will have levels assessed at T1 and T2, and supplementation will be given if initial levels are suboptimal. The control group will have levels assessed only at T2.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Dentistry, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in a de-identified format with other researchers, upon request, for further scientific investigation. The data sharing process will adhere to ethical guidelines and privacy laws to ensure participant confidentiality and security. All shared data will be anonymized, and no personally identifiable information will be included.
Supporting Information: SAP
Time Frame: Individual participant data (IPD) and supporting information will be available for sharing starting from February 20, 2025, and will remain accessible until November 25, 2025. During this time, researchers can request access to de-identified data for further scientific investigations.

REFERENCES:
- [Result] Al-Attar A, Abid M. The Effect of Vitamin D3 on the Alignment of Mandibular Anterior Teeth: A Randomized Controlled Clinical Trial. Int J Dent. 2022 Feb 14;2022:6555883. doi: 10.1155/2022/6555883. eCollection 2022. PMID 35198025